CLINICAL TRIAL: NCT07133243
Title: TESTI : Testicular Torsion Evaluation by ultraSonography Technic Imaging
Brief Title: Testicular Torsion Evaluation by ultraSonography Technic Imaging
Acronym: TESTI
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Roubaix (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-016
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Testicular Torsion
MeSH Terms: conditions — Spermatic Cord Torsion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single arm
  Interventions: Other: testicular ultrasound

INTERVENTIONS:
Other: testicular ultrasound — each patient will receive an testicular ultrasound to confirm diagnostic of testicular torsion

SUMMARY:
The goal of this observational study is to assess the diagnostic concordance between testicular Doppler ultrasound of the spermatic cord vessels performed by an emergency physician and the diagnosis of testicular torsion made by the urologist during an exploration in the operating room (Gold standard) in men patients between 16 to 70 years old with suspicion of testicular torsion.

Participants will receive ultrasound performed by emergency physician during their visit to the emergency department. Results of this exam will be compare to gold standard. If the results are consistent, the investigators will have demonstrated the value of integrating ultrasound by the emergency physician into the management of testicular torsion.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Minimum age of 16 years and maximum age of 70 years
* Presenting with unilateral testicular pain lasting less than 72 hours
* Admitted to the Roubaix Hospital Emergency
* Presence of an emergency physician trained in performing testicular ultrasound during the transition to the Emergency unit
* Patient who did not object to participating in the study

Exclusion Criteria:

* Recent history (less than one month) of ipsilateral testicular torsion, testicular trauma, or testicular surgery
* Patient with a history of sex reassignment, currently undergoing sex reassignment, or taking sex reassignment hormones
* Innate or acquired absence of one of the two testicles within the scrotum
* Patient who has already been included once in the TESTI study

Ages: 16 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population will be selected from male (from 16 to 70) presenting testicular pain in emergency unit of Roubaix's hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-03 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of patient with diagnostic of testicular torsion | At enrollement
  Concordance between testicular ultrasound and chirurgical diagnostic of testicular torsion

SECONDARY OUTCOMES:
Identify predictive factors for diasgnosis of testicular torsion | At enrollement
  Describe the predictive factors for the diagnosis of testicular torsion by multimodal regression including demographic data, clinical signs and complementary lab results.
Epidemiological factors of testicular pain | At enrollement
  Describe the epidemiological factors of testicular pain based on age and antedecents
Doppler result concordance between emergency physician and radiologist | From enrollement to 48 hours
  Compare the results between testicular ultrasound performed by an emergency physician and the same ultrasound performed by a radiologist
Characterised patients who benefit ultrasound from a radiologist according to final diagnostic | From enrollement to 48 hours
  Simple description of the demographic, epidemiological and clinical characteristics of patients who benefited from an ultrasound at 48 hours by a radiologist according to the final diagnosis retained

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Roubaix, Roubaix, France

IPD SHARING:
Plan to Share IPD: No